CLINICAL TRIAL: NCT05251493
Title: Intravenous Iron Isomaltoside Versus Iron Sucrose for Treatment of Iron Deficiency in Pregnancy: A Randomized Comparative Trial
Brief Title: Ferric Derisomaltose (Iron Isomaltoside) Versus Iron Sucrose for Treatment of Iron Deficiency in Pregnancy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Collaborators: Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Principal Investigator, Ryan Lett, Physician Lead Patient Blood Management Department, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC6-024-c260086 SHA REB-21-64
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency Anaemia in Childbirth
Keywords: quality of life; anemia
MeSH Terms: conditions — Anemia | interventions — iron isomaltoside 1000; ferric derisomaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Intervention Model Description: IDA is associated with poor neonatal outcomes and maternal morbidity. This clinical trial will compare IV iron isomaltoside to IV iron sucrose for correction of IDA, along with the potential impacts to the patient: physical, emotional and convenience of attending, receiving and follow up appointments associated with iron infusion. The study will also take into consideration the financial and resource impacts to the healthcare system, and to the patient, and determine the validity of using iron isomaltoside and iron sucrose in second and third trimester pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron Isomaltoside/ferric derisomaltose (Active Comparator): route: intravenous Dosage: 1000-1500 mg (100mg/mL), max dose 20mg/kg Frequency: max dose 1000 mg, if further doses required, must receive dosage divided Duration: one infusion or two infusions (dose dependent)
  Interventions: Drug: Iron Isomaltoside 1000, ferric derisomaltose
- Iron Sucrose (Active Comparator): Route: Intravenous Dosage: 100 mg/mL (maximum 300 mg per dose) Frequency: up to 3 doses per week or 1000 mg per week maximum Duration: until iron needs reached by simplified table
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron Isomaltoside 1000, ferric derisomaltose — iron isomaltoside 20 mg/mL
  Other Names: Monoferric DIN 22477777
  Arms: Iron Isomaltoside/ferric derisomaltose
Drug: Iron sucrose — iron sucrose 100 mg/mL
  Other Names: iron sucrose DIN 02502917
  Arms: Iron Sucrose

SUMMARY:
Ion deficiency anemia (IDA) is associated with poor neonatal outcomes and maternal morbidity. Iron replacement may be done with oral iron or intravenous iron, with intravenous iron being utilized later in pregnancy or if there is an inadequate response to oral iron in the first trimester. In Canada, iron sucrose has been used, however iron isomaltoside is as safe as other formulations of IV iron but can replete iron stores with a single visit. Replenishing iron stores reduces both maternal and neonatal risks and is supported by current guidelines. Iron status may play a role in depression, as well as anemia, bleeding and blood transfusion.

The goal of this clinical trial:

* Correct IDA with fewer visits and less impact on the healthcare system
* Improve the health and well being of all pregnant women who are experiencing moderate to severe iron deficiency anemia.

DETAILED DESCRIPTION:
IDA is associated with poor neonatal outcomes and maternal morbidity. This clinical trial will compare IV iron isomaltoside to IV iron sucrose for correction of IDA, along with the potential impacts to the patient: physical, emotional and convenience. The study will also take into consideration the financial and resource impacts to the healthcare system, as well as determine the validity of using iron isomaltoside in second and third trimester pregnancy.

The trial will be a randomized, comparative, single center, phase III trial with a 1:1 allocation ratio. There will be two groups involved in this trial. Group 1: A single dose of IV iron isomaltoside. Group 2: Standard iron sucrose therapy.

Eligible participants will be screened for IDA during the initial appointment (greater or equal to 13 weeks gestational age) with the obstetrical care provider. Discussion/awareness about the study will be discussed at their appointment or over the telephone with the obstetrical care provider. This information will only be discussed if the patient requires IV iron repletion in second or third trimester pregnancy.

Enrollment inclusion/exclusion criteria must be met for the participant to receive the information about the study.

Study personnel will discuss the clinical trial, including obtaining informed consent with the eligible participant. Baseline vital signs and blood work will be documented from the previous patient visit where IDA was diagnosed. Documentation and data collection will occur at 3 other points within the clinical trial: Post iron infusion (approximately 30 days after infusion), during delivery and at 6 weeks postpartum.

Standard community blood work requisitions will be used for blood work and blood tests that occur within the community or health clinic setting. Standard Physician orders or Pre Printed orders will be followed for tests, bloodwork and medication administration while in hospital at the delivery admission. Participant duration will be from intake (approximately 13 weeks gestation to 6 week follow up post delivery of infant). The follow up at the 6 week appointment will be the end point for the participation of the study. A total of approximately 231 days of involvement within the study duration for each participant.

The study will be completed 36 months after the enrollment of the first participant or when all patients have been recruited to satisfy the sample size calculation.

The sample size is calculated based on the primary endpoint (achievement of Hb≥110 g/L after iron intervention). As iron isomaltoside has a faster rise in hgb (weeks 1 to 5) with fewer visits, it is assumed that 5% of iron isomaltoside and 15% of iron sucrose participants will have hgb <110 g/L at delivery. Given the 10% difference between groups of patients achieving a hgb ≥110g/L in the iron isomaltoside group, it is calculated that at a p of 0.05 and a power of 80%, 140 participants are required in each treatment group.

The primary endpoint of this trial is the correction of anemia, defined as Hgb greater or equal to 110 g/L at trial post iron infusion (30 days post iron infusion (with measured hemoglobin levels during delivery and at six weeks postpartum).

The secondary endpoint is the change in quality of life questionnaires from baseline, post iron infusion, at delivery and 6 weeks postpartum through standard Redcap tools. Additionally, any adverse event will be documented with appropriate follow up care.

Participant subjective data will also be collected based on tolerance of IV iron, pregnancy related symptoms and quality of life comparing pre iron infusion, post iron infusion, at delivery and again at 6 weeks post delivery. Participants will also be required to answer questions related to convenience of appointment for iron infusion(s), accessibility to the infusion appointments and post birth bonding with baby.

Analysis will be performed after data collection is complete using the latest version of RStudio. Qualitative variables will be expressed as counts, percentages, quantitative variables as mean +/- standard deviation or median (interquartile range [IQR] depending on the variable distribution. Comparison of continuous variables will be performed using the two sided Student's t test or Mann Whitney U test (where appropriate), and the chi squared test or Fisher's exact test (where appropriate) to compare category variables. The Kaplan Meier method will be used for the graphical assessment of time related events. Analysis of the primary efficacy and safety endpoints will be by intention to treat.

Participants who withdraw either due to medical condition or expressed withdrawal will be set as censored. No data relating to the withdrawal will be utilized in the data analysis. The proportion of endpoints will be analyzed using logistic regression. Continuous secondary endpoints will be analyzed by linear regression. For analyzing missing data, model based multiple imputations will be used for both primary and secondary outcomes.

Eligible pregnant women with iron deficiency will be recruited through the Department of Obstetrics and Gynecology Department, or through health care providers that maintain obstetrical care privileges at RGH.

Treatments arms will be allocated through a blocked randomization list prepared by an online tool. Moreover, the randomization will be stratified by Hgb level in increments of 10g/L to pursue equal distribution of the two groups. The sequence list will not be accessible to the investigators. Participants will be randomly assigned to receive either IV iron isomaltoside or IV iron sucrose. IV iron sucrose is the comparator because it is currently the formulation used for IDA during second and third trimester pregnancy in Regina, Saskatchewan, Canada. Products will be stored as per the product monograph and as per requirements and guidelines set out by the Saskatchewan Health Authority.

The Saskatchewan Health Authority will ensure that the written agreement to perform trial related monitoring, audits, Research Ethics Board reviews and regulatory inspections, and provide direct access to source data and/or documents of this clinical trial, as required. Data and source documents must be readily available to the Research Ethics Board, Health Canada, Therapeutic Products Directorate, inspectors, clinical trial team members, including investigators and/or obstetrical care providers for the purposes of compliance with regulatory requirements of the clinical protocol and purposes relating to treatment, care and follow up of adverse drug reactions or by means of trace back/lookback as required. Source data and documentation include patient records whether hard copy or electronic, blood work, appointment dates and times, test and procedure results relating to this clinical trial. All source documents must be accessible during the clinical trial period and after the clinical trial has completed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* Pregnancy with Gestational age ≥13 weeks
* Iron deficiency anemia defined as:
* Hemoglobin less than or equal to 110g/L and
* Serum ferritin less than 30ng/mL or
* Iron Saturation (Iron/TIBC) less than 20%
* Willing to participate and attend all planned follow up visits
* Willing to sign informed consent form
* Willing to attend appointments for iron infusion and follow up visits
* Willing to attend all planned bloodwork appointments

Exclusion Criteria:

* Pregnancy GA less than 13 weeks
* History of anemia caused by thalassemia or other haematologic disorder other than iron deficiency anemia ,
* Known serious hypersensitivity to other parental iron products
* Iron overload or disturbances in utilization of iron (i.e, haemochromatosis and haemosiderosis)
* Decompensated liver cirrhosis or active hepatitis
* History of multiple allergies
* Active acute or chronic infections
* Treated with IV iron products or blood transfusion within 4 weeks prior to inclusion
* Current participation in any other interventional trial
* Multiple gestation pregnancy
* Significant comorbidities (asthma requiring daily therapy or other lung diseases)
* Heart disease
* Kidney disease
* Rheumatologic disease
* Cancer
* Known hypersensitivity to iron sucrose or any excipients
* Known hypersensitivity to iron isomaltoside or any excipients.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females with diagnosed iron deficiency anemia
Enrollment: 280 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Correction of anemia | 30 days post iron infusion
  defined as (hemoglobin) hgb greater or equal to 110 g/L (grams per litre) for all participants
Correction of anemia | at delivery admission
  defined as (hemoglobin) hgb greater or equal to 110 g/L (grams per litre), all participants of clinical trial
Correction of anemia | 6 week post partum visit
  defined as (hemoglobin) hgb greater or equal to 110 g/L (grams per litre), all participants

SECONDARY OUTCOMES:
Participant's tolerance to IV iron infusion | Collected at delivery admission survey
  Tolerance of IV (intravenous) iron infusion (assigned arm)-subjective data collection/ collection of data for adverse events if applicable/ All participants
Comparison of participant's pregnancy related symptoms- subjective measure | collected from baseline, at delivery and 6 weeks postpartum
  Measure of pregnancy related symptoms from each point in the clinical trial -subjective data collection/ All participants
Convenience/barriers of IV iron appointment(s)- subjective measure | collected at delivery admission, post iron infusion
  Measure of participant's convenience of appointment and barriers to accessing the IV iron- subjective data collection
Changes in Participant's Mental Health and Physical Well-Being | baseline (at intake), post iron infusion (1 week after infusion), at delivery, at 6 weeks post partum
  Comparison of participant's physical and mental well being changes across the span of the study- subjective data collection for all participants
Reported bonding with baby-subjective | collected at 6 weeks postpartum
  Participant's reported post birth bonding with baby. (subjective data collection for all participants)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lett, MD, FRCPC, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavord S, Daru J, Prasannan N, Robinson S, Stanworth S, Girling J; BSH Committee. UK guidelines on the management of iron deficiency in pregnancy. Br J Haematol. 2020 Mar;188(6):819-830. doi: 10.1111/bjh.16221. Epub 2019 Oct 2. No abstract available. PMID 31578718
- [Background] Wesstrom J. Safety of intravenous iron isomaltoside for iron deficiency and iron deficiency anemia in pregnancy. Arch Gynecol Obstet. 2020 May;301(5):1127-1131. doi: 10.1007/s00404-020-05509-2. Epub 2020 Apr 8. PMID 32270330
- [Background] Congdon EL, Westerlund A, Algarin CR, Peirano PD, Gregas M, Lozoff B, Nelson CA. Iron deficiency in infancy is associated with altered neural correlates of recognition memory at 10 years. J Pediatr. 2012 Jun;160(6):1027-33. doi: 10.1016/j.jpeds.2011.12.011. Epub 2012 Jan 11. PMID 22244466
- [Background] Pollock RF, Muduma G. A budget impact analysis of parenteral iron treatments for iron deficiency anemia in the UK: reduced resource utilization with iron isomaltoside 1000. Clinicoecon Outcomes Res. 2017 Aug 10;9:475-483. doi: 10.2147/CEOR.S139525. eCollection 2017. PMID 28848355
- [Background] Holm C, Thomsen LL, Norgaard A, Langhoff-Roos J. Single-dose intravenous iron infusion or oral iron for treatment of fatigue after postpartum haemorrhage: a randomized controlled trial. Vox Sang. 2017 Apr;112(3):219-228. doi: 10.1111/vox.12477. Epub 2017 Feb 15. PMID 28198084
- [Background] Khalafallah AA, Dennis AE, Ogden K, Robertson I, Charlton RH, Bellette JM, Shady JL, Blesingk N, Ball M. Three-year follow-up of a randomised clinical trial of intravenous versus oral iron for anaemia in pregnancy. BMJ Open. 2012 Oct 18;2(5):e000998. doi: 10.1136/bmjopen-2012-000998. Print 2012. PMID 23087011
- [Background] Diagnostic and Statistical Manual of Mental Disorders: DSM-5. 5th ed., American Psychiatric Association, 2013. doi.org.db29.linccweb.org/10.1176/ appi.
- [Background] Duley L, Uhm S, Oliver S; Preterm Birth Priority Setting Partnership Steering Group. Top 15 UK research priorities for preterm birth. Lancet. 2014 Jun 14;383(9934):2041-2042. doi: 10.1016/S0140-6736(14)60989-2. No abstract available. PMID 24931684